CLINICAL TRIAL: NCT02134847
Title: Multi-center Clinical Trial of Limiting Resident Work Hours on ICU Patient Safety
Acronym: ROSTERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christopher P. Landrigan, MD, MPH, Dr., Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2010P001346
Record Dates: First submitted 2013-03-15; First posted 2014-05-09 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Physician Fatigue
Keywords: Resident; Fatigue; Sleep deprivation; medical errors
MeSH Terms: conditions — Fatigue; Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention cohort (Experimental): This cohort will work on the SCS intervention schedule
  Interventions: Other: SCS intervention schedule
- Control cohort (No Intervention): This group will work on a traditional schedule

INTERVENTIONS:
Other: SCS intervention schedule
  Arms: Intervention cohort

SUMMARY:
In this proposal, we seek to address conclusively two knowledge gaps: 1) the lack of data on the relationship between PGY2+ (post graduate year 2) sleep deprivation and patient safety; and 2) the lack of data on the relationship between resident sleep deprivation and preventable patient injuries. Through the Clinical and Translational Science Award (CTSA)-funded Sleep Research Network, the largest and only federally-funded sleep science network in the U.S., we propose conducting a multi-center randomized crossover trial in six pediatric ICUs staffed by PGY2 and PGY3 residents. We will compare rates of all serious errors (i.e., rates of harmful and other serious medical errors due to any cause, including but not limited to fatigue-related errors, handoff errors, and provider knowledge deficits) of a sleep and circadian science-based (SCS) intervention schedule with a traditional schedule that includes frequent shifts of 24 hours or longer. Our specific aims will be:

1. To test the hypothesis that PGY2&3 residents working on an SCS intervention schedule will make significantly fewer harmful medical errors (preventable adverse events) and other serious medical errors (near misses) while caring for ICU patients than residents working on a traditional schedule; (primary endpoints: resident-related preventable adverse events and near misses)
2. To test the hypothesis that rates of harmful medical errors (preventable adverse events) and other serious medical errors (near misses) throughout the ICU (i.e., those involving and those not involving residents) will be lower in ICUs when PGY2&3 residents work on an SCS intervention schedule than when residents work on a traditional schedule; (major secondary endpoints: ICU-wide preventable adverse events and near misses)
3. To test the hypothesis that resident physicians' risk of neurobehavioral performance failures and motor vehicle crashes - as assessed through simple visual reaction time tasks [Johns Drowsiness Score (JDS) and Psychomotor Vigilance Task (PVT) lapses] - will be lower on the SCS intervention schedule than on the traditional schedule. (major secondary endpoints: resident neurobehavioral performance and predicted driving safety)

ELIGIBILITY:
Inclusion Criteria:

* Must be a second or third year resident of pediatrics or a combined pediatrics program

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-03-05 (Actual); Study Completion 2017-03-05 (Actual)

PRIMARY OUTCOMES:
resident-related preventable adverse events and near misses. | Each resident (subject) will be observed for 1 month.
  PGY2&3 residents working on an SCS intervention schedule will make significantly fewer harmful medical errors (preventable adverse events) and other serious medical errors (near misses) while caring for ICU patients than residents working on a traditional schedule;(primary endpoints: resident-related preventable adverse events and near misses)

SECONDARY OUTCOMES:
ICU-wide preventable adverse events and near misses | Each participating PICU will be studied for 8 months on each of the schedules (16 months total).
  Rates of harmful medical errors (preventable adverse events) and other serious medical errors (near misses) throughout the ICU (i.e., those involving and those not involving residents) will be lower in ICUs when PGY2&3 residents work on an SCS intervention schedule than when residents work on a traditional schedule.
resident neurobehavioral performance. | Subjects will be tested 3-5 times per week for 1 month.
  Resident physicians' risk of neurobehavioral performance failures as assessed through simple visual reaction time tasks [Psychomotor Vigilance Task (PVT) lapses] - will be lower on the SCS intervention schedule than on the traditional schedule.
Risk of resident motor vehicle crashes (MVC) | Subjects will be monitored while they drive to/from work for 1 month.
  Fatigue during the commute to and from work, as assessed by the John's drowsiness scale (JDS), will be lower on the SCS schedule than the traditional schedule, making MVC's less likely during the time on the SCS schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Landrigan, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Charles A Czeisler, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (6):
- United States (6):
  - Childrens Hospital of Colorado, Aurora, Colorado
  - University of Iowa Hospital, Iowa City, Iowa
  - Childrens Hospital Boston, Boston, Massachusetts
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - University of Virginia Health System, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Rahman SA, Sullivan JP, Barger LK, St Hilaire MA, O'Brien CS, Stone KL, Phillips AJK, Klerman EB, Qadri S, Wright KP Jr, Halbower AC, Segar JL, McGuire JK, Vitiello MV, de la Iglesia HO, Poynter SE, Yu PL, Sanderson AL, Zee PC, Landrigan CP, Czeisler CA, Lockley SW; ROSTERS STUDY GROUP. Extended Work Shifts and Neurobehavioral Performance in Resident-Physicians. Pediatrics. 2021 Mar;147(3):e2020009936. doi: 10.1542/peds.2020-009936. Epub 2021 Feb 22. PMID 33619044
- [Derived] Landrigan CP, Rahman SA, Sullivan JP, Vittinghoff E, Barger LK, Sanderson AL, Wright KP Jr, O'Brien CS, Qadri S, St Hilaire MA, Halbower AC, Segar JL, McGuire JK, Vitiello MV, de la Iglesia HO, Poynter SE, Yu PL, Zee PC, Lockley SW, Stone KL, Czeisler CA; ROSTERS Study Group. Effect on Patient Safety of a Resident Physician Schedule without 24-Hour Shifts. N Engl J Med. 2020 Jun 25;382(26):2514-2523. doi: 10.1056/NEJMoa1900669. PMID 32579812
- [Derived] Barger LK, Sullivan JP, Blackwell T, O'Brien CS, St Hilaire MA, Rahman SA, Phillips AJK, Qadri S, Wright KP, Segar JL, McGuire JK, Vitiello MV, de la Iglesia HO, Poynter SE, Yu PL, Zee P, Sanderson AL, Halbower AC, Lockley SW, Landrigan CP, Stone KL, Czeisler CA; ROSTERS Study Group. Effects on resident work hours, sleep duration, and work experience in a randomized order safety trial evaluating resident-physician schedules (ROSTERS). Sleep. 2019 Aug 1;42(8):zsz110. doi: 10.1093/sleep/zsz110. PMID 31106381
- [Derived] Blackwell T, Kriesel DR, Vittinghoff E, O'Brien CS, Sullivan JP, Viyaran NC, Rahman SA, Lockley SW, Barger LK, Halbower AC, Poynter SE, Wright KP Jr, Yu PL, Zee PC, Landrigan CP, Czeisler CA, Stone KL; ROSTERS Study Group. Design and recruitment of the randomized order safety trial evaluating resident-physician schedules (ROSTERS) study. Contemp Clin Trials. 2019 May;80:22-33. doi: 10.1016/j.cct.2019.03.005. Epub 2019 Mar 15. PMID 30885799

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT02134847/Prot_SAP_000.pdf